CLINICAL TRIAL: NCT02027493
Title: Safety and Efficacy of Hansenula-Derived Pegylated-Interferon Alpha-2a and Ribavirin Customized Combination Therapy in Egyptian Children With Chronic Hepatitis C Infection
Brief Title: Hansenula-Derived Pegylated-Interferon Alpha-2a in Egyptian Children With Chronic HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Collaborators: Yassin Abdelghaffar Charity Center for Liver Disease and Research (Other); National Hepatology & Tropical Medicine Research Institute (Other Government); Ain Shams University (Other); Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa M. Sira, Associate Professor of Pediatric Hepatology, National Liver Institute, Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLI-YAGCC-CUPH-HCV-PEG-PED
Record Dates: First submitted 2014-01-01; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Children; Chronic hepatitis C; Hansenula polymorpha; Pegylated interferon; Response rate; Ribavirin; Treatment
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reiferon R weekly plus ribavirin (Active Comparator): patients who continued treatment on weekly basis (7-day schedule). This group included patients who were HCV-RNA negative at week 12 and those who had < 1 log decrease in HCV-RNA viremia
  Interventions: Drug: Reiferon R; Drug: Ribavirin
- Reiferon R (every 5-day) plus ribavirin (Active Comparator): patients who continued treatment on a 5-day schedule. This group included patients who had ≥ 1 log decrease in viremia (compared to pre-treatment level) at week 12
  Interventions: Drug: Reiferon R; Drug: Ribavirin

INTERVENTIONS:
Drug: Reiferon R — subcutaneous injection of 100 μg/m2
  Other Names: Hansenula-derived pegylated interferon alpha 2a; Reiferon Retard
Drug: Ribavirin — 15 mg/kg daily on two divided doses

SUMMARY:
Egypt has the highest prevalence of hepatitis C virus infection in adults (up to 20%) and children (up to 5.5%). The major genotype (90%) is type 4. Pegylated interferon-alpha-2a or -2b and ribavirin have been used in small numbers of hepatitis C virus-infected children with sustained virological response being higher in genotypes 2 and 3 than in genotypes 1 and 4. Genotype 4 is has been described as difficult-to-treat genotype. Several attempts to modify treatment protocols have been tried in adults in an attempt to achieve higher rates of sustained virological response. Shortening injection interval and/or treatment duration prolongation have been tried with variable outcome reports.

A novel Hansenula- derived pegylated interferon alpha 2a: 20 Kilo dalton (Reiferon Retard) has been used over the last 4 years in the Egyptian market.

We aimed to investigate the safety and efficacy of Reiferon retard plus ribavirin customized regimen in hepatitis C virus-RNA seropositive Egyptian children. Forty six children with chronic hepatitis C virus aged 3-19 years were selected from 3 hepatic tertiary centers.

Clinical and laboratory evaluation were undertaken. Quantitative polymerase chain reaction (PCR) for HCV-RNA was done before starting treatment, at 4, 12, 24, 48, 72 weeks during treatment and 6 months after stoppage of treatment. All patients were assigned to receive a weekly subcutaneous injection of pegylated interferon alpha 2-a ( Reiferon Retard) plus oral Ribavirin daily for 12 weeks ,then cases were divided according to PCR results into 2 groups.

Group I: Patients who continued treatment on weekly basis: this group included patients who had negative PCR at week 12 as well those who had positive PCR without any change in viremia. Group II: Patients who continued treatment on a 5- days schedule: this group included patients who had any decrease in viremia at week 12.

Patients who were PCR-negative at week 48 and had at least one PCR-positive test during therapy were assigned to have an extended treatment course of 6 months duration.

The occurrence of adverse effects was assessed during treatment and follow up

DETAILED DESCRIPTION:
hepatitis C virus is a major health problem, not only in adults but also in the pediatric age group. In Egypt, the prevalent genotype is the difficult-to-treat genotype 4. Attempts are being made to improve the treatment outcomes. In the current study we aim to investigate the effect of customized pegylated interferon-alpha-2a plus ribavirin in children with chronic hepatitis C virus. For that, 46 children with chronic hepatitis C virus were recruited from three tertiary Pediatric Hepatology centers. All were assigned to receive weekly subcutaneous pegylated interferon-alpha-2a plus daily ribavirin for 12 weeks. At this point, the study population was divided into two arms. Arm 1 included those who became hepatitis C virus-RNA negative by polymerase chain reaction and those who showed no change of viremia or a decrease of less than 1 log. This group continued treatment on weekly bases for 48 weeks, even those who are hepatitis C virus-RNA positive. Arm 2; included patients who had a decrease in viremia more than one log of pre-treatment viremia level. For those patients, injection interval was shortened to every 5-day for a completion period of 48 weeks. Patients from either group who were polymerase chain reaction-negative at week 48, but had at least one polymerase chain reaction-positive test during therapy, were assigned to have an extended treatment course up to 72 weeks.

So the first customization was,

1. prolongation of treatment duration for up to 48 weeks regardless response type
2. Shortening injection interval in some patients to every 5-day injection
3. The third customization was the prolongation of treatment for extra 6 months, i.e. up tp 72 weeks in some patients.

The occurrence of adverse effects, virological and biochemical responses were assessed during treatment and follow up.

ELIGIBILITY:
Inclusion Criteria:

* children aged 3-19 years
* compensated chronic HCV infection (HCV-RNA positive by PCR for more than 6 months)
* whose hemoglobin was ≥10 g/dL
* neutrophilic count > 1500/mm3
* platelet count > 75,000/mm3
* normal random blood sugar
* normal serum creatinine
* normal serum ferritin
* normal thyroid function tests
* normal lipid profile
* no other causes of liver disease (autoimmune hepatitis, Wilson disease, alpha one antitrypsin deficiency nor hepatitis B virus infection).
* Liver biopsy was mandatory for enrollment

Exclusion Criteria:

* decompensated cirrhosis
* any other cause of liver disease associating HCV infection
* body mass index ≥ 95 percentile
* severe psychiatric conditions
* uncontrolled seizure disorder
* decompensated cardiovascular disease, renal insufficiency
* evidence of retinopathy
* decompensated thyroid disease
* hemoglobinopathy
* immunologically mediated diseases or any other chronic illness requiring long term immunosuppressive drugs
* previous interferon therapy within one year of enrollment

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To study the safety of Hansenula-Derived Pegylated-Interferon Alpha-2a (Reiferon retard) in attaining sustained virological response in children with chronic hepatitis C virus infection | 48 weeks
  The efficacy and Safety was assessed during the 48 weeks of therapy, patients were monitored clinically, laboratory for the appearance of any side effects

SECONDARY OUTCOMES:
Efficacy of treatment customization on the outcome | 96 weeks
  To assess the effect of tailoring treatment [by decreasing the interval between injection (5days vs 7 days) and prolonging duration of therapy (48 weeks vs 72 weeks)] on sustained virological response based on the on-treatment virologic response

OTHER OUTCOMES:
To assess predictors of sustained virological response | 96 weeks
  1. compare demographic parameters in responders and non-responders
  2. comparing pretreatment hepatitis C viremia in responders and non-responders
  3. compare expected duration of infection in responders and non-responders
  4. compare histopathological changes in responders and non-responders
  5. compare pretreatment liver enzymes in responders and non-responders
  6. compare treatment duration in responders and non-responders
  7. compare injection interval in responders and non-responders

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M Sira, M.D., Study Director — Pediatric Hepatology Department, National Liver Institute, Menofiya University, Shebin El-koom, 32511 Menofiya, Egypt; Tawhida Y Abdel-Ghaffar, M.D., Principal Investigator — Yassin Abdel Ghaffar Charity Center for Liver Disease and Research, 2851 Cairo, Egypt; Suzan El Naghi, M.D., Study Director — Pediatric Department, National Hepatology and Tropical Medicine Research Institute, 11441 Cairo, Egypt; Hanaa El-Karaksy, M.D., Study Chair — Cairo University; Heba Helmy, M.D., Study Chair — Cairo University; Mona S El-Raziky, M.D., Study Chair — Cairo University; Elham F Abdel-Aty, M.Sc., Study Chair — Pediatric Hepatology Department, National Liver Institute, Menofiya University, Shebin El-koom, 32511 Menofiya, Egypt; Aleef A Allam, M.D., Study Chair — Pediatric Hepatology Department, National Liver Institute, Menofiya University, Shebin El-koom, 32511 Menofiya, Egypt; Hanaa A El-Araby, M.D., Study Chair — Pediatric Hepatology Department, National Liver Institute, Menofiya University, Shebin El-koom, 32511 Menofiya, Egypt; Behairy E Behairy, M.D., Study Chair — Pediatric Hepatology Department, National Liver Institute, Menofiya University, Shebin El-koom, 32511 Menofiya, Egypt; Mohamed A El Guindi, M.D.; Ph.D., Study Chair — Pediatric Hepatology Department, National Liver Institute, Menofiya University, Shebin El-koom, 32511 Menofiya, Egypt; Hatem El-Sebaie, M.D., Study Chair — Biochemistry Department, National Liver Institute, 32511 Menofiya, Egypt; Aisha Y Abdel-Ghaffar, M.D., Study Chair — Clinical Pathology Department, Ain Shams University, Cairo, Egypt; Nermin A Ehsan, M.D., Study Chair — Pathology Department, National Liver Institute, Menofiya University, Shebin El-koom, 32511 Menofiya, Egypt; Ahmad El-Hennawy, M.D., Study Chair — Pathology Department, Cairo University, Faculty of Medicine, Kasr El-Aini, Cairo, Egypt
Locations (3):
- Egypt (3):
  - Department of Pediatrics, Cairo University Pediatric Hospital, Cairo, Cairo Governorate
  - National Liver Institute, Menoufiya, Menofiya
  - Yassin Abdel Ghaffar Charity Center for Liver Disease and Research, Cairo

REFERENCES:
- [Derived] El Naghi S, Abdel-Ghaffar TY, El-Karaksy H, Abdel-Aty EF, El-Raziky MS, Allam AA, Helmy H, El-Araby HA, Behairy BE, El-Guindi MA, El-Sebaie H, Abdel-Ghaffar AY, Ehsan NA, El-Hennawy AM, Sira MM. Safety and efficacy of Hansenula-derived PEGylated-interferon alpha-2a and ribavirin combination in chronic hepatitis C Egyptian children. World J Gastroenterol. 2014 Apr 28;20(16):4681-91. doi: 10.3748/wjg.v20.i16.4681. PMID 24782620